CLINICAL TRIAL: NCT02856620
Title: The Role of Cardiac Mechanics, Circulating Biomarkers and Frailty in Aortic Stenosis in Predicting Outcomes After Aortic Valve Intervention.
Brief Title: The Role of Cardiac Mechanics, Biomarkers and Frailty in Aortic Stenosis
Acronym: SCRABLES
Status: Recruiting | Type: Observational
Sponsor: Christine Henri (Other)
Responsible Party: Sponsor-Investigator, Christine Henri, Assistant Professor of Medicine, Montreal Heart Institute
Organization: Montreal Heart Institute (Other)
Other Study IDs: MontrealHI
Record Dates: First submitted 2016-07-26; First posted 2016-08-05 (Estimated); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure; Aortic Stenosis
Keywords: cardiac mechanics; circulating biomarkers; frailty
MeSH Terms: conditions — Heart Failure; Aortic Valve Stenosis; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — NT-proBNP hs-TnT sST2 hs-CRP GDF-15
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Moderate AS with HF
  Interventions: Other: Observational only
- Severe AS with HF
  Interventions: Other: Observational only
- Moderate AS without HF
  Interventions: Other: Observational only
- Severe AS without HF
  Interventions: Other: Observational only
- HFpEF without AS
  Interventions: Other: Observational only
- Normal age-matched controls
  Interventions: Other: Observational only

INTERVENTIONS:
Other: Observational only — Observational only

SUMMARY:
The role of cardiac mechanics, circulating biomarkers and frailty in predicting outcomes in patients with aortic stenosis after aortic valve replacement (SCRABLES -The 2-Parts Study) Part I: Observational study to characterize phenotypes, structural alterations and biomarkers profiles in a broad spectrum of patients with aortic stenosis and heart failure with preserved ejection fraction (HFpEF).

Part II: Prospective cohort study to characterize patients' phenotypes, cardiac structural alterations, circulating biomarkers and frailty in order to optimize risk stratification and patient selection for aortic valve intervention.

DETAILED DESCRIPTION:
Part I: This part will be an observational exploratory analysis to collate available data from Treatment of preserved cardiac function heart failure with an aldosterone antagonist trial (TOPCAT) cohort regarding the potential role of clinical phenotype, structural alterations and biomarkers profiles that can help determine symptom severity in a AS and HFpEF, and offer insights into which patients with AS may suffer from HFpEF after aortic valve replacement (AVR).

Part II: This part will be a prospective cohort study to create an AS functional capacity score that will include phenotypic classification, structural alterations using novel echocardiographic parameters such as cardiac mechanics, biomarkers profiles and frailty evaluation in order to more accurately predict functional capacity before (Segment A) and after aortic valve intervention (Segment B) and to compare with healthy control group (Segment C).

ELIGIBILITY:
Inclusion Criteria:

Part I - Patients part of the TOPCAT cohort from Americas fulfilling inclusion criteria of Part II-Group 3 (see below) and/or patients enrolled in the Part II study

Part II - Segment A and B Age ≥ 18 years old AS classified according to aortic valve area measured by Doppler echocardiography Group 1: Moderate AS (1.0-1.5cm2) Group 2: Severe AS (1cm2) Group 3: HF with preserved left ventricular ejection fraction (LVEF ≥45%) without significant AS

Part II - Segment C (Control Group) Age ≥ 18 years old Healthy subject taking into account exclusions parameters at the time of screening Able to sign the consent form

Exclusion Criteria:

Part I and II - Segment A and B Prior AVR either by surgery or trans-aortic valve implantation; Severe mitral valve disease or aortic regurgitation; LVEF < 45% Myocardial infarction within the previous 3 months; Angina limiting the 6MWTD and thought to be the result of severe coronary artery disease; Cerebrovascular transient ischemic attack or stroke within the previous 6 months; Known active infection or cancer; renal insufficiency (glomerular filtration rate <30 mL/min/1.73m2) or end-stage renal disease; Significant anemia (haemoglobin <90 g/L) or thrombocytopenia (platelet count <50), history of bleeding diathesis or coagulopathy; Life expectancy <12 months due to non-cardiac co-morbid conditions; Chronic obstructive pulmonary disease with Global initiative for chronic obstructive lung disease (GOLD) stages 3-4; musculoskeletal disease limiting the ability to perform the 6MWTD.

Part II - Segment C (Control Group) History of cardiovascular disease Risk factors associated with cardiovascular (treated diabetes, hypertension, body mass index >30kg/m2) Pregnancy or breastfeeding All other cause from Segment A and B

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Part I: The study population will be recruited from the TOPCAT cohort and Part -II.
  Part II: Patients will be recruited from cardiology, heart failure, TAVI and cardiac surgery clinics, echocardiography laboratory of the MHI and as for the control group from publicity in and out of the MHI.
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2016-07; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
6-Minutes Walk Test Distance (6MWTD) | 12 to 18 months

SECONDARY OUTCOMES:
Kansas City Cardiomyopathy Questionnaire (KCCQ) | 12 to 18 months
The Physical Ability Score (PAS) | 12 to 18 months
Occurrence of major adverse events defined as stroke, myocardial infarction, pacemaker implantation, prolonged (>14 days) or re-hospitalization, lack of reduction in doses of diuretics, new onset of heart failure and mortality | 12 to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Christine Henri, MD, Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No